CLINICAL TRIAL: NCT04343092
Title: Effectiveness of Ivermectin as add-on Therapy in COVID-19 Management (An Externally Controlled Pilot Trial)
Brief Title: Effectiveness of Ivermectin as add-on Therapy in COVID-19 Management
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Faiq Gorial, Professor and consultant rheumatologist, University of Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO20040001
Record Dates: First submitted 2020-04-05; First posted 2020-04-13 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ivermectin (IVM)+ Hydroxychloroquin (HCQ)+ Azithromycin (AZT) (Experimental): Ivermectin 12 mg /weekly )+ Hydroxychloroquine 400mg/daily + azithromycin 500mg daily
  Interventions: Drug: Ivermectin (IVM)

INTERVENTIONS:
Drug: Ivermectin (IVM) — Ivermectin 0.2 mg /kg (single dose at once =2 tablets of 6mg/weekly
  Other Names: Ivermectin

SUMMARY:
Comparing the effectiveness of Ivermectin( IVM) +Hydroxychloroquin + azithromycin (AZT) group to Hydroxychloroquin (HCQ) + azithromycin (AZT)

DETAILED DESCRIPTION:
Comparing effectiveness of single dose 0.2mg/kg Ivermectin (IVM) plus hydroxychloroquine (HCQ) 400mg BID in first day then 200mg BID for 5 days plus azithromycin (AZT) 500mg in first day then 250mg for 5 days.

The comparison group was a historical control population and data collected from the current study were compared to that historical control population

ELIGIBILITY:
Inclusion Criteria:

-1. Patients with age above 18 years and any gender with definite Dx of covid19 and pneumonia in the ward according to the clinical, laboratory, and imaging criteria.

2. Understands and agrees to comply with planned study procedures.

Exclusion Criteria:

1. Patients with hypersensitivity or severe adverse effects to Ivermectin
2. Renal impairment
3. Hepatic impairment.
4. Pregnancy or a desire to become pregnant (drug considered pregnancy category c)
5. Breast feeding.
6. Patient with covid 19 positive and mild no pneumonia
7. Children under the age of five or those who weigh less than 15 kilograms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-04-18 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faiq I Gorial, Professor, Principal Investigator — University of Baghdad; Jawad I. Rasheed, Study Chair — Arab Board for Health Specialiazation in Iraq
Locations (1):
- General Directorate of Medical City, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ivermectin (IVM)+ Hydroxychloroquin (HCQ)+ Azithromycin (AZT)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ivermectin (IVM)+ Hydroxychloroquin (HCQ)+ Azithromycin (AZT): IVM 0.2mg /kg single dose at admisison day HCQ 400mg BID in the first day then 200mg BID for 5 days AZT 500mg in the first day then 250mg for 5 days
Arm/Group | Ivermectin (IVM)+ Hydroxychloroquin (HCQ)+ Azithromycin (AZT)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.87 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Iraq | 16
Severity of CoVID-19 Symptoms [Count of Participants; unit: Participants] — Severity of COVID-19 were measured according to WHO criteria for grading COVID-19
  Participants
    Mild | 9
    moderate | 7
Clinical features [Count of Participants; unit: Participants]
  Cough | 13
  Fever | 11
  Shortness of breath | 9
  Myalgia | 8
  Sore throat | 4
Comorbidity ( underlying diseases) [Number; unit: participants]
  Diabetes melitus | 3
  Hypertension | 3
  Asthma | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Cured Patients
Description: Primary outcome is assessed by calculating the number of patients who had symptoms free and two successive readings of negative PCR swab.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Groups:
- IVM+HCQ+AZT Group: Time to cure in IVM+HCQ+AZT group and evaluated by measuring time from admission of the patient to the hospital till discharge after being free of symptoms and negative PCR swab. Once nasopharyngeal and oropharyngeal swab viral PCR testing yielded negative results 2 times consecutively, no further testing was performed.
Arm/Group | IVM+HCQ+AZT Group
Number analyzed (Participants) | 16
Participants | 16

2. Secondary Outcome: Time to Cure of COVID-19 Patients in the IVM +HCQ+AZT Group
Description: Time to cure is evaluated by measuring time from admission of the patient to the hospital till discharge after being free of symptoms and negative PCR swab. Once nasopharyngeal and oropharyngeal swab viral PCR testing yielded negative results 2 times consecutively, no further testing was performed
Time Frame: 4 week
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | IVM+HCQ+AZT Group
Number analyzed (Participants) | 16
Days | 7.62 (2.75)
Statistical Analysis 1: Comparison: IVM+HCQ+AZT Group; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 7.92; Historical control population included: Hydroxychloroquin (HCQ) 400mg BID at admission day then 200mg BID for 5 days plus Azithromycin (AZT) 500mg at admission day then 250mg for 5 days

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- IVM+HCQ+AZT Group: Assessment of any adverse events in 0.2mg IVM single dose on admission day +HCQ 400mg BID in the first day then 200mg BID for 5 days+AZT 500mg in the first day then 250mg for 5 days
Arm/Group | IVM+HCQ+AZT Group
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
small sample size; single center design, and short time for the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT04343092/Prot_SAP_000.pdf